The GlaxoSmithKline group of companies

 Division
 : Worldwide Development

 Information Type
 : Reporting and Analysis Plan (RAP)

Title : Reporting and Analysis Plan for a Randomized double blind (sponsor unblind) study evaluating the effect of 14 days of treatment with danirixin (GSK1325756) on neutrophil extracellular traps (NETs) formation in participants with stable chronic obstructive pulmonary disease (COPD)

Compound Number : GSK1325756

Effective Date : 14-NOV-2018

### **Description:**

• The purpose of this RAP is to describe planned efficacy and safety analyses and output to be included in the Clinical Study Report (CSR) for Protocol 207551.

• This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverable.

### **RAP Author(s):**

| Approver | Date | Approval Method |
|---|---|---|
| Statistician (Respiratory Clinical Statistics) | 13-NOV-2018 | e-mail |
| Programming Manager (Respiratory Clinical Programming) | 14-NOV-2018 | e-mail |

Copyright 2018 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

## The GlaxoSmithKline group of companies

## **RAP Team Approvals:**

| Approver | Date | Approval Method |
|---------------------------------------------|-------------|-----------------|
| PPD CONT. | 13-NOV-2018 | e-mail |
| Physician (CIL) | | |
| Principal Clinical Research Scientist (OSL) | 13-NOV-2018 | e-mail |
| PPD PPD | | |
| Principal Data Manager (DQL) | 13-NOV-2018 | e-mail |

## **Clinical Statistics and Clinical Programming Line Approvals:**

| Approver | Date | Approval Method |
|---|---|---|
| Project Statistician (Respiratory Clinical Statistics) On behalf of PPD Line Manager (Respiratory Clinical Statistics) | 14-NOV-2018 | e-Signature |
| Project Programmer (Respiratory Clinical Statistics) On behalf of PPD Line Manager (Respiratory Clinical Statistics) | 14-NOV-2018 | e-Signature |

## **TABLE OF CONTENTS**

| | | | | PAGE |
|---|---|---|---|---|
| 1. | INTR | ODUCTIO | ON | 6 |
| 2 | CLIM | MADV OF | F KEY PROTOCOL INFORMATION | 0 |
| 2. | | | | |
| | 2.1. | Change | es to the Protocol Defined Statistical Analysis Plan | 5 |
| | 2.2. | | Objective(s) and Endpoint(s) | |
| | 2.3. | | Design | |
| | 2.4. | Statistic | cal Hypotheses / Statistical Analyses | 8 |
| 3. | PI AN | INFD AN | ALYSES | q |
| Ο. | 3.1. | | Analyses | |
| | 3.2. | | nalyses | |
| | | | • | |
| 4. | | | PPULATIONS | |
| | 4.1. | Protoco | ol Deviations | 10 |
| 5. | CONS | SIDERAT | TIONS FOR DATA ANALYSES AND DATA HANDLING | |
| ٥. | | | 18 | 12 |
| | 5.1. | | Freatment & Sub-group Display Descriptors | |
| | 5.2. | | ne Definitions | |
| | 5.3. | | nation of Covariates, Other Strata and Subgroups | |
| | | 5.3.1. | Covariates and Other Strata | |
| | 5.4. | Multiple | e Comparisons and Multiplicity | 13 |
| | 5.5. | Other C | Considerations for Data Analyses and Data Handling | |
| | | Conver | ntions | 13 |
| _ | ОТШ | W DODLI | ILATION ANALYOFO | 4.4 |
| 6. | 6.1. | | LATION ANALYSESew of Planned Study Population Analyses | |
| | 0.1. | Overvie | ew of Flatified Study Fopulation Arialyses | 14 |
| 7. | EFFI( | CACY AN | IALYSES | 15 |
| | 7.1. | | y Efficacy Analyses | |
| | | 7.1.1. | | |
| | | 7.1.2. | · | |
| | | 7.1.3. | | |
| | | 7.1.4. | Strategy for Intercurrent (Post-Randomization) Events | 15 |
| | | 7.1.5. | Statistical Analyses / Methods | |
| | | | 7.1.5.1. Statistical Methodology Specification | |
| | 7.2. | Second | dary Efficacy Analyses | |
| | | 7.2.1. | Endpoint / Variables | |
| | | 7.2.2. | Summary Measure | 16 |
| | | 7.2.3. | Population of Interest | |
| | | 7.2.4. | Statistical Analyses / Methods | |
| | | 7.2.5. | Endpoint / Variables | |
| | | 7.2.6. | Summary Measure | |
| | | 7.2.7. | Population of Interest | |
| | | 7.2.8. | Statistical Analyses / Methods | |
| | | | 7.2.8.1. Statistical Methodology Specification | |
| | 7.3. | Explora | atory Efficacy Analyses | |
| | | 7.3.1. | Éndpoint / Variables | |

| 8. | SAFE | TY ANALY | /SES | | 19 |
|---|---|---|---|---|---|
| | 8.1. | | | alyses | |
| | 8.2. | | | Special Interest Analyses | |
| | 8.3. | | | Analyses | |
| | 8.4. | Other Sa | ifety Analys | es | 19 |
| 9. | PHAR | MACOKIN | IETIC ANA | LYSES | 20 |
| ٠. | 9.1. | | | inetic Analyses | |
| | | 9.1.1. | | Variables | |
| | | | | Drug Concentration Measures | |
| | | | | Derived Pharmacokinetic Parameters | |
| 10. | POPU | LATION F | PHARMACO | OKINETIC (POPPK) ANALYSES | 21 |
| 11. | REFEI | RENCES. | | | 22 |
| 12 | APPFI | NDICES | | | 23 |
| | 12.1. | Appendix | k 1: Protoco | ol Deviation Management and Definitions for Per | |
| | | Protocol | Population. | | 23 |
| | | 12.1.1. | Exclusions | s from Per Protocol Population | 23 |
| | 12.2. | Appendix | k 2: Schedu | lle of Activities | 24 |
| | | | | efined Schedule of Events | |
| | 12.3. | | | ment Windows | |
| | | | | of Assessment Windows for Analyses | 26 |
| | 12.4. | Appendix<br>Events | k 4: Study F | Phases and Treatment Emergent Adverse | 27 |
| | | 12.4.1. | | ses | |
| | | 12.1.1. | | Study Phases for Concomitant Medication | |
| | | 12.4.2. | | Emergent Flag for Adverse Events | |
| | 12.5. | | k 5: Data Di | splay Standards & Handling Conventions | 28 |
| | | 12.5.1. | | Process | |
| | | 12.5.2. | | Standards | |
| | | 12.5.3. | | Standards for Pharmacokinetic | |
| | 12.6. | Appendix | | l and Transformed Data | |
| | | 12.6.2. | Study Pop | ulation | 30 |
| | | 12.6.3. | Efficacy | | 31 |
| | | 12.6.4. | Dataset to | Protocol Mapping | 31 |
| | 12.7. | Appendix | 7: Reporti | ng Standards for Missing Data | 33 |
| | | 12.7.1. | | · Withdrawals | |
| | | 12.7.2. | Handling of | of Missing Data | 33 |
| | | | | Handling of Missing and Partial Dates | |
| | 12.8. | Appendix | k 8: Values | of Potential Clinical Importance | 34 |
| | | 12.8.1. | Laboratory | / Values | 34 |
| | | 12.8.2. | | | |
| | | 12.8.3. | | S | |
| | 12.9. | | | tion Pharmacokinetic (PopPK) Analyses | 36 |
| | | 12.9.1. | | n Pharmacokinetic (PopPK) Dataset | |
| | | | • | on | 36 |
| | | | 12.9.1.1. | 3 3 1 | |
| | | | 10015 | Data | 36 |
| | | | 12.9.1.2. | Handling Missing Dose Times | 36 |

207551

| | | 12.9.1.3. H | landling Missing Times of PK Samples | 36 |
|---|---|---|---|---|
| | | 12.9.1.4. H | landling of PK Data Below the Lower Limit of | |
| | | | Quantification | |
| | | 12.9.1.5. D | ataset Specification | 36 |
| 12.10. | Appendix | 10: Abbrevia | ations & Trade Marks | 48 |
| | 12.10.1. | Abbreviation | S | 48 |
| | 12.10.2. | Trademarks | | 49 |
| 12.11. | Appendix | 11: List of D | ata Displays | 50 |
| | 12.11.1. | Data Display | Numbering | 50 |
| | 12.11.2. | Mock Examp | ole Shell Referencing | 50 |
| | 12.11.4. | Study Popula | ation Tables | 51 |
| | | | les | |
| | 12.11.6. | Efficacy Figu | ıres | 56 |
| | | | S | |
| | 12.11.8. | Pharmacokir | netic Tables | 61 |
| | 12.11.9. | Pharmacokir | netic Figures | 62 |
| | 12.11.10 | <b>ICH Listings</b> | | 64 |
| | | | tings | |
| 12.12. | | | e Mock Shells for Data Displays | |

## 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol

| Revision Chronology | | |
|---------------------|-------------|----------|
| 2017N314013_00 | 16-MAY-2017 | Original |

## 2. SUMMARY OF KEY PROTOCOL INFORMATION

## 2.1. Changes to the Protocol Defined Statistical Analysis Plan

| Protocol | Protocol Reporting & Analysis Plan | |
|---|---|---|
| Statistical Analysis Plan | Statistical Analysis Plan | Rationale for Changes |
| <ul> <li>Enrolled - All participants<br/>who sign informed<br/>consent</li> </ul> | Enrolled - All participants who sign informed consent and for whom a record exists on the study database | Align with standard Enrolled population definition. |
| Randomised | <ul> <li>mITT population<br/>defined to be used for<br/>selected displays</li> </ul> | Used for key displays |
| Primary completer | <ul> <li>Population definition<br/>refined</li> </ul> | To allow for missing data and increase clarity |
| • Safety | mITT population used for safety reporting | Safety population not required. |
| <ul> <li>PK population</li> </ul> | <ul> <li>PK population defined</li> </ul> | Used for PK displays |
| <ul> <li>Endpoint - Model specific<br/>PK parameters of danirixin<br/>(e.g., oral clearance, oral<br/>steady state volume of<br/>distribution).</li> </ul> | Danirixin concentration<br>and standard<br>pharmacokinetic (PK)<br>parameters for<br>danirixin (e.g. AUC,<br>Cmax, tmax) | Updated due to small number of participants with PK data |
| <ul> <li>Endpoints - serum IL-8 or<br/>sputum mucin</li> </ul> | Removed | Not collected |
| Primary analysis Bayesian | Primary analysis Frequentist | The primary analysis has been simplified as the historical data could not be used as a prior. |
| <ul> <li>Modified Primary<br/>Completer</li> </ul> | Population defined | Defined to allow for a sensitivity<br>around the definitions of quality for<br>the samples |

# 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To assess the change from<br>baseline in NETs formation in<br>participants with COPD following<br>14 days of treatment with danirixin<br>hydrobromide (HBr) 35mg twice<br>daily | Reduction in sputum NETs (quantified by Histone-<br>elastase complexes) |
| Secondary Objectives | Secondary Endpoints |
| To assess the change from<br>baseline in NETs formation in<br>participants with COPD following<br>14 days of treatment with danirixin<br>HBr 35mg twice daily | <ul> <li>Reduction in sputum NETS (quantified by Deoxyribonucleic acid [DNA]-elastase complexes)</li> <li>Reduction in sputum NET area quantification by microscopy</li> </ul> |
| To further characterize the safety<br>of danirixin HBr 35mg tablets<br>compared with placebo in<br>participants with COPD | <ul><li>Adverse events</li><li>Vital Signs</li><li>ECG</li><li>Spirometry</li></ul> |
| To assess the effects of danirixin<br>HBr 35mg twice daily on NETosis-<br>associated biomarkers in sputum<br>and peripheral blood | <ul> <li>Change from baseline in sputum resistin levels</li> <li>Change from baseline in the ratio of sputum NETs to sputum neutrophils</li> <li>Change from baseline in sputum elastase activity</li> <li>Change from baseline in peripheral blood neutrophil NET formation (DNA release)</li> </ul> |
| Characterise the population pharmacokinetic (PK) profile of approximately 14 days of dosing of danirixin HBr 35mg twice daily in participants with COPD | Danirixin concentration and standard pharmacokinetic (PK) parameters for danirixin (e.g. AUC, Cmax, tmax) |
| Exploratory Objectives | Exploratory Endpoints |
| To explore the relationships<br>between NETs formation and lung<br>microbiome composition | Characterize sputum microbiome composition and diversity |
| To explore volatile organic compound (VOC) profile in participants with COPD | <ul> <li>Characterize relationship between lung microbiome and exhaled volatile organic compounds (VOCs) in stable COPD</li> <li>To explore variability of exhaled VOCs</li> </ul> |
| To explore the effects of danirixin | Changes from baseline in ex-vivo neutrophil |

| Objectives | Endpoints |
|---|---|
| HBr 35mg twice daily on | phagocytosis of bacteria by flow cytometry |
| neutrophil activity and exploratory biomarkers | <ul> <li>Changes in exploratory urine, sputum and blood<br/>biomarkers (e.g. plasma fibrinogen, serum C-<br/>reactive protein)</li> </ul> |

## 2.3. Study Design



## 2.4. Statistical Hypotheses / Statistical Analyses

The objective of this study is to assess whether danirixin impacts NET formation in participants with COPD. There will be no formal hypotheses tests and significant tests. Model based results for the primary endpoint of reduction in sputum NETs (quantified by Histone-elastase complexes) adjusted for baselin, will be used.

## 3. PLANNED ANALYSES

## 3.1. Interim Analyses

There is no formal interim analysis planned for this study. Although, blinded data looks were performed at 12 participants and 19 participants. The purpose of the data looks is to check data quality. The data showed that 6 participants had poor quality data. The team decided to replace all 6 participants; approximately 30 participants will be enrolled.

## 3.2. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. After decision to terminate DNX in COPD the study was stopped early. 19 subjects had completed the study.
- 2. All required database cleaning activities have been completed and final database release (DBR)
- 3. All criteria for unblinding the randomization codes have been met.
- 4. Randomization codes have been distributed according to RandAll NG procedures.
- 5. Database freeze (DBF) has been declared by Data Management.

## 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Enrolled | | |
| whom a record exists on the study database. This population will be used for the tables/listings of reasons for withdrawal before randomization and listings of AEs and SAEs for non-randomized | | Reasons for<br>withdrawal before<br>randomization. |
| | participants. | <ul> <li>Inclusion, exclusion,<br/>and randomization<br/>criteria deviations</li> </ul> |
| Modified ITT | | |
| one dose of study treatment. Participants will be analysed according to the treatment they actually | | Efficacy |
| | received. If a participant received more than one treatment during the treatment period, they will be reported according to the treatment taken the most based on doses taken from each container. | Safety |
| Primary | All participants in the Modified ITT population who | Sputum NETs |
| Completer | have completed the assessments supporting the primary endpoint (sputum NETs). • In the case where the modified ITT and the primary completer population are the | Secondary NETs analyses |

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| | same, the primary completer population will not be defined and all output will be done on the Modified ITT population. • Participants need sputum samples of acceptable quality at screening/baseline and day 14. • Acceptable quality samples have viable leukocytes >50% and coded as acceptable or good in MISPQL | |
| Modified Primary<br>Completer | All participants in the Modified ITT population who have completed the assessments supporting the primary endpoint (sputum NETs). • In the case where the modified ITT and the primary completer population are the same, the primary completer population will not be defined and all output will be done on the Modified ITT population. • Participants need sputum samples of reasonable quality at screening/baseline and day 14. Reasonable quality samples have viable leukocytes >50% and coded as acceptable, good or poor quality in MISPQL This population will only be use if this increases the available sample from the Primary completer population by 20%. | Secondary NETs<br>analyses |
| PK | All participants in the mITT population who had at least 1 non-missing PK assessment (Non-quantifiable [NQ] values will be considered as non-missing values) obtained and analysed whilst on treatment with danirixin. | • PK |

**NOTES:** Please refer to Appendix 11: List of Data Displays which details the population to be used for each displays being generated.

### 4.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan 17Aug2017 Final V1.0.

o Data will be reviewed prior to freezing the database to ensure all important deviations are captured and categorised on the protocol deviations dataset.

• This dataset will be the basis for the summaries and listings of protocol deviations.

A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

## 5.1. Study Treatment & Sub-group Display Descriptors

| Treatment Group Descriptions | | | |
|---|---|---|---|
| RandAll NG System Data Displays for Reporting | | | |
| Code | Description | Description | Order in TLF |
| PBO | Placebo | Placebo | 1 |
| DNX | GSK1325756 (danirixin) 35mg | DNX 35mg BD | 2 |
| | HBr | _ | |

Treatment comparisons will be displayed as follows using the descriptors as specified:

1. Danirixin vs. Placebo

## 5.2. Baseline Definitions

| Parameter | Study Assessments Conside | Baseline Used in<br>Data Display | |
|---|---|---|---|
| | Screening (Visit 0 / Visit 1) | Day 1 (Visit 2) | |
| Induced sputum variables | X | X | Baseline |
| Vital signs | | X | Baseline |
| Spirometry variables | | X | Baseline |
| ECG [mean of triplicate] | | X | Baseline |
| Clinical Laboratory Assessments | | X | Baseline |

For labs, vitals and ECG, use the most recent value prior to dosing. In cases where the induced sputum from day 1 does not meet quality standards, the sample from screening can be used.

## 5.3. Examination of Covariates, Other Strata and Subgroups

#### 5.3.1. Covariates and Other Strata

Other covariates will be included for specific analyses as detailed in model specifications in Section 7.1 and Section 7.2.

| Category | Details |
|------------|---------------------|
| Covariates | Treatment, baseline |

## 5.4. Multiple Comparisons and Multiplicity

No adjustment for multiplicity is required for this study, as the primary analysis involves an estimation approach, rather than hypothesis testing.

# 5.5. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---------|----------------------------------------------------------------|
| 12.3 | Appendix 3: Assessment Windows |
| 12.4 | Appendix 4: Study Phases and Treatment Emergent Adverse Events |
| 12.5 | Appendix 5: Data Display Standards & Handling Conventions |
| 12.6 | Appendix 6: Derived and Transformed Data |
| 12.7 | Appendix 7: Reporting Standards for Missing Data |
| 12.8 | Appendix 8: Values of Potential Clinical Importance |

## 6. STUDY POPULATION ANALYSES

## 6.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the modified ITT population, unless otherwise specified.

Study population analyses including analyses of subject's disposition, protocol deviations, demographic and baseline characteristics, prior and concomitant medications, and exposure and treatment compliance will be based on GSK Core Data Standards. Details of the planned displays are presented in Appendix 11: List of Data Displays.

#### 7. EFFICACY ANALYSES

## 7.1. Primary Efficacy Analyses

#### 7.1.1. Endpoint / Variables

The primary endpoint will be the percent change (relative to baseline) in sputum NETs, quantified by Histone-elastase complexes, for danirixin.

#### 7.1.2. Summary Measure

Mean and 95% confidence interval will be calculated for the danirixin and placebo arms at day 7 and 14.

## 7.1.3. Population of Interest

The primary efficacy analysis will be based on the Primary Completer population, unless the primary completer populations is the same as the mITT population. In that case the mITT population will be used for all analysis. Participants with poor quality sputum samples should also be excluded from the analysis.

## 7.1.4. Strategy for Intercurrent (Post-Randomization) Events

No intercurrent events are considered of interest in this analysis. Data for the endpoint will be complete for the specific population

#### 7.1.5. Statistical Analyses / Methods

Unless otherwise specified, endpoints / variables defined in Section 7.1.1 will be summarised using descriptive statistics, graphically presented and listed.

#### 7.1.5.1. Statistical Methodology Specification

#### **Endpoint / Variables**

Sputum NETs quantified by Histone-elastase complexes

#### **Model Specification**

- The ratio of post-baseline NETs values to baseline NETS values will be log transformed prior to analysis. Note:  $\log\left(\frac{NETs_{post}}{NETs_{baseline}}\right) = \log\left(NETs_{post}\right) \log(NETs_{baseline})$ .
- $y_{ij} = \beta_{baselins} \cdot \log(x_i) + \beta_{treatment} \cdot x_i + \beta_{day \times treatment} \cdot x_{ij} + \gamma_i + \epsilon_{ij}$
- Where i is the index for each participant and j is the index for day

#### **Model Checking & Diagnostics**

- The mixed effect model will control for treatment, baseline, and day.
- An unstructured symmetric covariance structure will be used. Although if there are issues with convergence auto-regressive lag 1 can be used.
- It may be necessary to exclude placebo data from the analysis due to small cell size.
- The Kenward and Rodger method for approximating the denominator degrees of freedom and

correcting for bias in the estimated variance-covariance of the fixed effects will be used
 If there are any departure from the distributional assumptions, alternative models will be explored using appropriate transformed data. Residual plots will be checked.

#### **Model Results Presentation**

Refer to Appendix 12 for detailed description of tables, figures, and listings

### 7.2. Secondary Efficacy Analyses

#### 7.2.1. Endpoint / Variables

The endpoint will be the change (relative to baseline) in sputum NETs, quantified by DNA-elastase and microscopy sputum resistin levels, ratio of sputum NETs to sputum neutrophils, sputum neutrophils, and sputum elastase activity. The mapping to dataset values are as follows. NETs quantified by microscopy are mean percent NETs per field. For a mapping of protocol variables to dataset variables (see <u>Dataset to Protocol Mapping</u>)

#### 7.2.2. Summary Measure

Unadjusted mean and standard error will be calculated for the danirixin and placebo arms at baseline, day 7 and 14. Unadjusted mean and standard error will be calculated for the percent change from baseline and absolute change from baseline for danirixin and placebo arms at day 7 and 14.

#### 7.2.3. Population of Interest

Same as above, for NETs quantified by histone-elastase.

## 7.2.4. Statistical Analyses / Methods

Unadjusted means and standard errors will be calculated.

#### 7.2.5. Endpoint / Variables

Change from baseline in peripheral blood neutrophil NET formation.

#### 7.2.6. Summary Measure

Unadjusted mean and standard error will be calculated for the danirixin and placebo arms at baseline, day 7 and 14. Unadjusted mean and standard error will be calculated for the percent change from baseline danirixin and placebo arms at day 7 and 14

#### 7.2.7. Population of Interest

The mITT population will be used.

#### 7.2.8. Statistical Analyses / Methods

### 7.2.8.1. Statistical Methodology Specification

Unadjusted means and standard errors will be calculated.

## 7.3. Exploratory Efficacy Analyses

## 7.3.1. Endpoint / Variables

Exploratory endpoints include volatile organic compounds (VOC), ex-vivo neutrophil phagocytosis of bacteria by flow cytometry, and blood biomarkers. The blood biomarkers are plasma fibrinogen, serum C-reactive protein. Only VOCs from Cyranose, ex-vivo neutrophil phagocytosis and blood biomarkers will be part of SAC. No formal statistical analysis will be used to summarize the blood biomarkers, only unadjusted means. The urine will be stored for a two-year period, during which if there is a biomarker assay that comes forth that will support danirixin development program, analysis may be run.

The between tube, within day, and between day variability of the Cyaronose device will calculated using a multilevel multivariate model. Day will be the top level, followed by time of day, and tube. An unstructured covariance should be used to model the relationship between sensors, but the same covariance structure should be used across all tubes. Assume a constant variance between morning and afternoon and between days. Below is the model diagram for a single subject.



 $Y_{ijkl} = \mu + S_i + D_{i(j)} + T_{k(ij)} + \varepsilon_{ijkl}$ 

In the case where the multilevel multivariate model does not converge then treat each sensor as independent and just run the multilevel model. If the multilevel models do not coverage, day and time of day can be collapsed into a single time level, in which we will only provide the variability of time rather than within day and between day.

Sputum microbiome, VOCs, and the relationship there in, will be investigated, but not included in the SAC due to the length of time needed to analysed the microbiome. The sputum microbiome will be analysed by Dundee. A secondary RAP to investigate VOCs and sputum microbiome will be written by the Computational Biology group to detail the analysis for this data. The results of this analysis will be written up in a report and added as an addendum to the CPSR.

#### 8. SAFETY ANALYSES

The safety analyses will be based on the mITT population.

#### 8.1. Adverse Events Analyses

Adverse events analyses including the analysis of adverse events (AEs), Serious (SAEs) and other significant AEs will be based on GSK Core Data Standards. The details of the planned displays are provided in Appendix 11: List of Data Displays.

## 8.2. Adverse Events of Special Interest Analyses

A comprehensive list of MedDRA terms based on clinical review will be used to identify each type of event. SRT, safety review team, has decided the Infective Pneumonia SMQ will used to identify AESI. The details of the planned displays are provided in Appendix 11: List of Data Displays.

## 8.3. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of Chemistry laboratory tests, Haematology laboratory tests, Urinalysis, and liver function tests will be based on GSK Core Data Standards. The details of the planned displays are in Appendix 11: List of Data Displays. The blood biomarkers, plasma fibrinogen and serum C-reactive protein, will be in the efficacy outputs.

## 8.4. Other Safety Analyses

The analyses of non-laboratory safety test results including ECGs and vital signs will be based on GSK Core Data Standards, unless otherwise specified. The details of the planned displays are presented in Appendix 11: List of Data Displays. Summaries of spirometry will also be created.

#### 9. PHARMACOKINETIC ANALYSES

#### 9.1. Primary Pharmacokinetic Analyses

#### 9.1.1. Endpoint / Variables

#### 9.1.1.1. Drug Concentration Measures

Refer to Appendix 5: Data Display Standards & Handling Conventions (Section 12.5.3 Reporting Standards for Pharmacokinetic)

#### 9.1.1.2. Derived Pharmacokinetic Parameters

Pharmacokinetic parameters will be calculated by standard non-compartmental analysis per current working practices and using the currently supported version of WinNonlin. All calculations of non-compartmental parameters will be based on actual sampling times. The pharmacokinetic parameters listed below will be determined from the blood concentration-time data on Day 1 and Day 14, as data permits.

| Parameter | Parameter Description |
|---|---|
| AUC(0-t) | Area under the concentration-time curve from time zero to the time of the last quantifiable concentration (C(t)) will be calculated using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid. |
| Cmax* | Maximum observed concentration, determined directly from the concentration-time data. |
| tmax | Time to reach Cmax, determined directly from the concentration-time data. |
| tlast | Time of last quantifiable concentration |

#### NOTES:

Additional parameters may be included as required.

Unless otherwise specified, endpoints / variables defined in Section 9.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

# 10. POPULATION PHARMACOKINETIC (POPPK) ANALYSES

PK data from this study may be combined with historic data for the purposes of population PK modelling which would be the subject of a separate analysis plan and would be presented separately from the main clinical study report (CSR).

To support this analysis a PopPK dataset will be generated. The details for the dataset specifications are provided in Section 12.8 Appendix 9.

## 11. REFERENCES

GlaxoSmithKline Document Number 2017N314013\_00, Protocol: Randomized double blind (sponsor unblind) study evaluating the effect of 14 days of treatment with danirixin (GSK1325756) on neutrophil extracellular traps (NETs) formation in participants with stable chronic obstructive pulmonary disease (COPD), 16 May 2017

## 12. APPENDICES

# 12.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population

## 12.1.1. Exclusions from Per Protocol Population

No per protocol analysis is defined in this study.

## 12.2. Appendix 2: Schedule of Activities

## 12.2.1. Protocol Defined Schedule of Events

Table 1 Schedule of activities

| Procedure | Pre-Screening and Screening <sup>1</sup> | | Treatment Period<br>(14 days) | | | Follow-up<br>Phone call | Unscheduled visit <sup>2</sup> | Notes |
|---|---|---|---|---|---|---|---|---|
| | V0 | V1 | V2 | V3 | V 4 | V5 | | |
| Day | Day -30 | to -1 | D 1 | D 7 | D14 | D 21 | As required | |
| Assessment window | | | | ±1d | ±1d | ±3d | As required | |
| Written, informed consent | Χ | | | | | | | |
| Inclusion and exclusion criteria | Χ | | | | | | | Recheck clinical status before randomization. |
| Demography, Medical history | Χ | | | | | | | |
| Baseline COPD assessment test (CAT) score | Х | | | | | | | |
| Adverse event (AE)/Serious adverse event (SAE) review | Χ | ←=======→ | | Х | X | | | |
| Concomitant medication review | Χ | + | -==== | ====== | $\rightarrow$ | Х | X | |
| Full physical examination including height and weight | Χ | | | | | | Х | |
| Vital signs | Χ | Х | Х | Х | Х | | Х | |
| Volatile organic compound (VOC) measurement | <b>X</b> 3 | X3,4 | <b>X</b> 5 | <b>X</b> 3 | <b>X</b> 3 | | Х | |
| Spirometry | Χ | | Х | | Х | | Х | |
| Induced Sputum Samples (including biomarker samples) | Χ | X 4 | Х | Х | Х | | Х | |
| Spirometry post-Sputum Induction | Χ | X 4 | Х | Х | Х | | Х | |
| Triplicate 12-lead ECG | | Х | Х | | Х | | Х | |
| Chest X-ray (historical within 1 year acceptable) | | Х | | | | | | |
| HIV, Hepatitis B and C screening | X6 | | | | | | | |
| Laboratory assessments (clinical chemistry including liver chemistries, haematology, biomarkers) | | X | | | Х | | Х | |
| Pharmacokinetic (PK) sample | | | | X8 | <b>X</b> <sup>7</sup> | | Х | See footnotes for timings of PK sampling |
| Genetic sample | | X9 | | | | | Pre-dose (baseline) sample. | |
| Urinary Pregnancy test (WOCBP only) | | X <sup>10</sup> | X <sup>10</sup> | | X <sup>10</sup> | | X <sup>10</sup> | |

| Procedure | Pre-Screening and Screening <sup>1</sup> | | Treatment Period<br>(14 days) | | | Follow-up<br>Phone call | Unscheduled visit <sup>2</sup> | Notes |
|---|---|---|---|---|---|---|---|---|
| | V0 | V1 | V2 | V3 | V 4 | V5 | | |
| Urinalysis (including biomarker samples) | | Х | Х | | Х | | Х | |
| Randomization | | | Х | | | | | All baseline assessments at V2 should be completed prior to randomization |
| Study treatment | | | Х | $\leftarrow \rightarrow$ | Х | | | |
| Dispense study medication | | | Х | | | | | |
| Monitor IP compliance (via manual counting and App) | | | Х | Χ | Χ | | | Digital App monitoring to begin at V2 |
| Collect IP | | | | | Χ | | | |

- The timing and number of planned study assessments, including safety, pharmacokinetic, pharmacodynamic/biomarker or other assessments may be altered during the course of the study based on newly available data (e.g., to obtain data closer to the time of peak plasma concentrations) to ensure appropriate monitoring.
- Any changes in the timing or addition of time points for any planned study assessments must be documented and approved by the relevant study team member and then
  archived in the sponsor and site study files, but will not constitute a protocol amendment. The IRB/IEC will be informed of any safety issues that require alteration of the safety
  monitoring scheme or amendment of the Informed consent form (ICF).
- Safety assessments should be performed in the following order where applicable/ possible: vital signs, ECG measurements, blood samples and spirometry.
  - 1. Screening visit is split into pre-screening on visit 0 and screening on visit 1 although the visits may be performed on the same day. This is to a) enable participants to potentially have more than one attempt at sputum induction for meeting eligibility and b) to only collect minimal screening data for subjects who fail on the basis of the elevated NETs since that is the key inclusion criteria that may not be known from medical records.
  - 2. Unscheduled visits may be used to collect information related to adverse events, for follow up of any safety assessments, and also to complete assessments where participants were not able to perform these within the visit window for any reason. It is not necessary to carry out all of the assessments listed under an unscheduled visit at a single visit; the assessments performed should be driven by the need for the visit.
  - 3. VOC measurement should be undertaken prior to sputum induction at these visits.
  - 4. Sputum induction (and associated VOC measurement and safety spirometry) at visit 1 is only necessary if participant unable to give sample at visit 0. Where the participant is judged by the investigator to have a borderline sputum NETs level (<0.5 units/ml) at visit 0, they will be invited to give a second sputum sample on visit 1 to re-assess eligibility.
  - 5. VOC measurements should be undertaken at the following timepoints at this visits: prior to sputum induction, and 4 hours post dose
  - 6. Hepatitis B (HBsAg) and Hepatitis C (HepC antibody) testing is required. If testing otherwise performed within 3 months prior to the first dose of study treatment, testing at screening is not required. Hepatitis C Ribonucleic acid (RNA) testing is optional; however a confirmatory negative Hepatitis C RNA test must be obtained, to be able to enroll participants with positive Hepatitis C antibody due to prior resolved disease.
  - 7. At visits 2 and 4, PK samples should be collected at the following time-points: pre-dose, 0.5, 1, 2 and 4 hours post-dose.
  - 8. At visit 3 only a pre-dose PK sample should be collected.
  - 9. Agreeing to genetic sample consent is not required for overall study participation. Informed consent for genetic sample must be obtained prior to taking sample.
  - 10. Pregnancy testing only required for women of child bearing potential (WOCBP). A positive urine pregnancy test requires confirmation with a serum pregnancy t

## 12.3. Appendix 3: Assessment Windows

## 12.3.1. Definitions of Assessment Windows for Analyses

Use nominal time of assessment.

# 12.4. Appendix 4: Study Phases and Treatment Emergent Adverse Events

#### 12.4.1. Study Phases

Assessments and events will be classified according to the time of occurrence relative to treatment start date.

| Study Phase | Definition |
|---|---|
| Pre-Treatment | Date ≤ Study Treatment Start Date |
| On-Treatment | Study Treatment Start Date < Date ≤ Study Treatment Stop Date +1 |
| Post-Treatment | Date > Study Treatment Stop Date +1 |

#### 12.4.1.1. Study Phases for Concomitant Medication

| Study Phase | Definition |
|---|---|
| Prior | If medication end date is not missing and is before date of start of treatment |
| Concomitant | Any medication that is not a prior |

#### NOTES:

 Please refer to Appendix 7: Reporting Standards for Missing Data for handling of missing and partial dates for concomitant medication. Use the rules in this table if concomitant medication date is completely missing.

## 12.4.2. Treatment Emergent Flag for Adverse Events

| Flag | Definition |
|---|---|
| Treatment<br>Emergent | If AE onset date is on or after treatment start date & on or before treatment stop date. |
| | Study Treatment Start Date ≤ AE Start Date ≤ Study Treatment Stop Date +1 |

#### NOTES:

- If the study treatment stop date is missing, then the AE will be considered to be On-Treatment.
- Time of study treatment dosing and start/stop time of AEs should be considered, if collected.

# 12.5. Appendix 5: Data Display Standards & Handling Conventions

#### 12.5.1. Reporting Process

| Software | |
|---|---|
| The currently | The currently supported versions of SAS Studio 3.6 (Basic Edition) will be used. |
| Reporting Area | Reporting Area |
| HARP Server | :\\UK1SALX00175.CORPNET2.com |
| HARP Compound | : \arprod\gsk1325756 |
| Analysis Datasets | |
| Analysis datasets will be created according to Legacy GSK A&R dataset standards. | |
| Generation of RTF Files | |
| RTF files will be generated for final analysis outputs | |

#### 12.5.2. Reporting Standards

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location: https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics
- Do not include subject level listings or figures in the main body of the GSK Clinical Study Report. All subject level listings should be located in the modular appendices as ICH or non-ICH listings

#### **Formats**

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF or provided by vendor.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.
  - For NETs the individual data will be provided according to the appropriate level of precision for the listings.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days
    on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the participant's listings.

| Unscheduled Visits | Unscheduled Visits |
|---|---|
| Unscheduled visit | <ul> <li>Unscheduled visits will not be included in summary tables and/or figures.</li> </ul> |
| All unscheduled v | risits will be included in listings. |
| <b>Descriptive Summar</b> | Descriptive Summary Statistics |
| Continuous Data | Continuous Data Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | Categorical Data N, n, frequency, % |
| Graphical Displays | |
| Refer to IDSL Statistical Principals 7.01 to 7.13. | |

## 12.5.3. Reporting Standards for Pharmacokinetic

| Pharmacokinetic Con | centration Data |
|---|---|
| PC Windows Non-<br>Linear (WNL) File | PC WNL file (CSV format) for the non compartmental analysis by Clinical Pharmacology Modelling and Simulation function will be created according to GUI_51487 and PKONE document. Note: Concentration values will be imputed as per GUI_51487 |
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | Refer to IDSL PK Display Standards. Refer to IDSL Statistical Principle 6.06.1. Note: Concentration values will be imputed as per GUI_51487 for descriptive summary statistics/analysis and summarized graphical displays only. Additionally, include geometric mean and 90% CI for the summary of blood concentration data |
| NONMEM/Pop PK<br>File | Pop-PK file (CSV format) for the POP-PK analysis by Clinical Pharmacology Modelling and Simulation function will be created according to the data specification detailed in Appendix 9. |
| NONMEM/PK/PD<br>File | Not applicable. |
| Pharmacokinetic Para | ameter Derivation |
| PK Parameter to be<br>Derived by<br>Programmer | None. |
| Pharmacokinetic Parameter Data | |
| Is NQ impacted PK<br>Parameters Rule<br>Being Followed | No. |
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | Refer to IDSL PK Display Standards. |

### 12.6. Appendix 6: Derived and Transformed Data

#### 12.6.1. General

#### Multiple Measurements at One Analysis Time Point

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- If there are two values within a time window (as per Section 12.3.1) the value closest to the target day
  for that window will be used. If values are the same distance from the target, then the mean will be
  taken.
  - For NETs: If there are unscheduled visits between screening and visit 2 use the last unscheduled visit prior to visit 2.
- Participants having both High and Low values for Normal Ranges at any post-baseline visit for safety parameters will be counted in both the High and Low categories of "Any visit post-baseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

#### **Study Day**

- Calculated as the number of days from First Dose Date:
  - Ref Date = Missing → Stu
    - → Study Day = Missing
  - Ref Date < First Dose Date → Study Day = Ref Date First Dose Date</li>
  - Ref Data ≥ First Dose Date → Study Day = Ref Date (First Dose Date) + 1

## 12.6.2. Study Population

#### **Treatment Compliance**

Treatment compliance will be calculated based on the formula:

# Treatment Compliance = Number of Actual Doses / (Planned Treatment Duration in Days \* Frequency)

- Frequency is 2 for BID Treatment compliance could be greater than 100% if there are events of overdose.
- Planned Treatment Duration is defined as 14 days

#### **Extent of Exposure**

• Number of days of exposure to study drug will be calculated based on the formula:

Duration of Exposure in Days = Treatment Stop Date - (Treatment Start Date) + 1

#### Age

- Age will be calculated based off the date participants signed consent forms
- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
  - Any participant with a missing day will have this imputed as day '15'.
  - Any participant with a missing date and month will have this imputed as '30th June'.
- Birth date will be presented in listings as 'YYYY'.

#### **Smoking Status**

- If the last smoked date (SUSMLSDT) is missing and a partial date (SUSMLSD) is not missing, then the
  following imputation should be applied to the partial smoking date for use in the reclassification of
  smoking status calculation:
  - o '01' will be used for the day and 'Jan' will be used for the month.

## **Treatment Compliance**

 Former smokers will be reclassified as current smokers if screening date – last smoked date < 183 days.

## **12.6.3.** Efficacy

## **Change from Baseline**

Change from Baseline will be calculated based on the formula:

## Change from Baseline = Value – Value on day 1

 Use the most recent pre-dose value for baseline. In the case where there is a bad sample on day 1 use screening

## 12.6.4. Dataset to Protocol Mapping

| Protocol Variable | BICAT<br>(BIOMARK) | MITEST<br>(MICROSCOPY) | MITSTD<br>(MICROSCOPY) | SPECTYPE<br>(MICROSCOPY) |
|---|---|---|---|---|
| Reduction in sputum NET area quantification by microscopy | | AK005 | 26 | C13278 |
| Reduction in sputum NETs<br>(quantified by<br>Histone-elastase<br>complexes) | HISTELAS | | | C13278 |
| Reduction in sputum NETS (quantified by Deoxyribonucleic acid [DNA]-elastase complexes) | DNAELAS | | | C13278 |
| Change from baseline in sputum resistin levels | RESIST | | | C13278 |
| Change from baseline in the ratio of sputum NETs to sputum neutrophils | | AW002 | | C13278 |
| Change from baseline in sputum elastase activity | ELASTASE | | | C13278 |

| Protocol Variable | BICAT | MITEST | MITSTD | SPECTYPE |
|---|---|---|---|---|
| | (BIOMARK) | (MICROSCOPY) | (MICROSCOPY) | (MICROSCOPY) |
| Change from baseline in peripheral blood neutrophil NET formation (DNA release, microscopy) | | AK005 | 8 | C12434 |

## 12.7. Appendix 7: Reporting Standards for Missing Data

## 12.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Participant study completion (i.e. as specified in the protocol) was defined as those who have completed the assessments supporting the primary endpoint</li> <li>Withdrawn participants may be replaced in the study.</li> <li>All available data from participants who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified.</li> </ul> |

## 12.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: |
| | <ul> <li>These data will be indicated by the use of a "blank" in participant listing displays.</li> <li>Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be<br/>missing data and should be displayed as such.</li> </ul> |
| Outliers | Any participants excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

12.7.2.1. Handling of Missing and Partial Dates

| | nanding of Missing and Partial Dates |
|---|---|
| Element | Reporting Detail |
| General | Partial dates will be displayed as captured in participant listing displays. |
| Adverse<br>Events | <ul> <li>The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: <ul> <li>Missing Start Day: First of the month will be used unless this is before the start date of study treatment; in this case the study treatment start date will be used and hence the event is considered On-treatment as per Appendix 4: Study Phases and Treatment Emergent Adverse Events.</li> <li>Missing Stop Day: Last day of the month will be used, unless this is after the stop date of study treatment; in this case the study treatment stop date will be used.</li> </ul> </li> <li>Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing.</li> <li>If treatment phase for an AE is missing due to missing dates class as on-treatment</li> </ul> |
| Concomitant<br>Medications/<br>Medical<br>History | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> </li> <li>The recorded partial date will be displayed in listings.</li> </ul> |

## 12.8. Appendix 8: Values of Potential Clinical Importance

## 12.8.1. Laboratory Values

| Hematology Analyte (units) | Effect | COPD | Patients |
|----------------------------------------------|---------|-------|----------|
| | | Low | High |
| Platelet Count (x109/L) | | 0.90x | 1.10x |
| Red Blood Cell Count (x1012/L) | | 0.93x | 1.07x |
| White Blood Cell Count (x10 <sup>9</sup> /L) | | 0.70x | 1.60x |
| Homoglobin (g/l) | Males | 0.85x | 1.20x |
| Hemoglobin (g/L) | Females | 0.85x | 1.20x |
| Hamataarit (Datia of 1) | Males | 0.50x | 1.30x |
| Hematocrit (Ratio of 1) | Females | 0.50x | 1.30x |
| MCV (fL) | | 0.25x | 2.00x |
| MCH (pg) | | 0.85x | 1.20x |
| Neutrophils (10^9/L) | | <1.0 | >10 |
| Lymphocytes (10^9/L) | | <1.2 | >11.2 |
| Monocytes (10^9/L) | | <0.16 | >2.6 |
| Eosinophils (10^9/L) | | | >1.2 |
| Basophils (10^9/L) | | | >0.85 |

Note: Multipliers are identified by "x", otherwise actual comparison values are provided with units.

| Chemistry Analyte | Effect | COPD Patients | |
|---|---|---|---|
| | | Low | High |
| BUN (mmol/L) | | 0.70x | 1.60x |
| | | | 1.30x |
| Creatinine (μmol/L) | | | (or >27 μmol/L increase from baseline) |
| Glucose (mmol/L) | | | 1.20x |
| Sodium (mmol/L) | | 0.80x | 1.15x |
| Potassium (mmol/L) | | 0.75x | 1.30x |
| Calcium (mmol/L) | Males | 0.85x | 1.08x |
| | Females | <0.499 mmol/l | >1.7465 mmol/l |
| Total Protein (mg/dL) | | | 1.25x |

Note: Multipliers are identified by "x", otherwise actual comparison values are provided with units.

| Liver Function Test Analyte | Effect | PCI Range | Unit |
|-----------------------------|--------|------------|--------|
| ALT/SGPT | High | ≥ 3x ULN | U/L |
| AST/SGOT | High | ≥ 3x ULN | U/L |
| Alkaline Phosphatase | High | ≥ 2x ULN | U/L |
| Direct Bilirubin | High | ≥ 1.5x ULN | μmol/L |

## 12.8.2. ECG

| ECG Parameter | PCI Range | Unit |
|------------------------------------|--------------|------|
| Absolute QTc Interval (QTcB, QTcF) | <300 or >500 | msec |
| QT Interval | <300 or >500 | msec |
| PR Interval | <120 or >210 | msec |
| QRS Interval | <70 or >125 | msec |
| Heart Rate | <35 or >120 | bpm |

Values based on the mean of triplicate

## 12.8.3. Vital Signs

| Vital Sign Parameter | PCI Range | Unit |
|--------------------------|-------------|-----------------|
| Systolic Blood Pressure | <90 or >160 | mmHg |
| Diastolic Blood Pressure | <40 or >110 | mmHg |
| Heart Rate | <35 or >120 | bpm |
| Respiration Rate | <8 or >30 | breaths<br>/min |

## 12.9. Appendix 9: Population Pharmacokinetic (PopPK) Analyses

## 12.9.1. Population Pharmacokinetic (PopPK) Dataset Specification

#### 12.9.1.1. Handling Missing Demographic and Covariate Data

Missing demographic and covariate data will not be imputed.

#### 12.9.1.2. Handling Missing Dose Times

Missing dose time information will be handled on a case by case basis by imputing this information based on prior dosing times or based on recorded PK collection times. The details of these imputations will be described in the report.

#### 12.9.1.3. Handling Missing Times of PK Samples

Missing times for PK will be handled on a case by case basis by imputing this information based on the dose time and/or times of other PK. The details of these imputations will be described in the report.

#### 12.9.1.4. Handling of PK Data Below the Lower Limit of Quantification

Any PK data below the lower limit of quantification will be set to missing.

#### 12.9.1.5. Dataset Specification

General description and rules:

- Missing or unknown values in covariates, if not to be imputed, will be assigned -99.
- The dataset is sorted by STUD, SUBJID, DATE, CTIM, EVID descending.
- The data items (columns) in the analysis-ready data file will be provided the same order as follows.
- Non-quantifiable (NQ) concentration values will be included as detailed for the CONC variable
- Non-numerical concentration values (such as NS, NR, NA) will not be included.
- Placebo subjects will not be included.
- The dataset will be a comma delimited ASCII text file and will be named:
  - NM.compound.study.PK.v1.csv
  - O Where "compound" is the compound name (e.g. GSK1234567) and "study" is the study number (e.g. 207551).
| Variable | Label<br>(Variable<br>description) | Туре | Units | Missing value | Codes/Derivation/Notes |
|---|---|---|---|---|---|
| ID | NONMEM<br>subject<br>identifier | Integer | None | Never | Sequential subject identifier across study after data is sorted by STUD, SUBJID, DATE, RTFD, EVID. Numbering to start at 1. To be entered in all rows for each subject. |
| STUDYID | Unique identifier for a study | Char | None | Never | 207551 for all records |
| STUD | Study ID | Num | None | Never | 207551 for all records |
| SUBJID | Subject<br>identifier for<br>study | Char | None | Never | Subject identifier, which must be unique within the study. The identification number of the subject as recorded on the CRF. Exclude placebo subjects. Include subjects who have received IP and have at least one measureable drug concentration. To be entered in all rows for each subject. |
| COUNTRY | Country | Char | None | Never | Country of the investigational site in which the subject participated in the trial; e.g. USA. To be entered in all rows for each subject. |
| SITEID | Unique identifier for a study site | Num | None | Never | e.g. PPD any lead zero should not be included. To be entered in all rows for each subject. |
| CONC | Drug<br>Concentration | Num | ng/mL | Never | CONC=0 for PK_GSK1325756 records. No sample (NS), insufficient sample (IS) and no result (NR) records will be excluded from dataset. CONC='.' for PK_GSK1325756 records < LOQ (i.e. if drug conc is NQ). |
| LNCONC | Natural log of CONC column | Num | ng/mL | Never | Natural log of CONC column. If CONC=0, then LNCONC='.'. |
| LLQ | Lower Limit of quantification | Num | ng/mL | Never | LLQ=5 or from source data if different. To be entered in all rows for each |

| Variable | Label<br>(Variable<br>description) | Туре | Units | Missing<br>value | Codes/Derivation/Notes |
|---|---|---|---|---|---|
| | | | | | subject. |
| LNLLQ | Natural log of LLQ column | Num | ng/mL | Never | Natural log of LLQ column. If LLQ=0, then LNLLQ='.'. |
| MATRIX | Sample matrix | Num | None | Never | MATRIX=1 (blood). |
| MATRTEXT | Sample matrix text | Char | None | Never | Text corresponding to code for MATRIX. Enter 'Blood' for all rows. |
| LABL | Label describing the record | Char | None | Never | LABL explains the type of measurement for CONC for the current record. LABL=DOSE_GSK1325756 for dose record. LABL=PK_GSK1325756 for blood concentration record. |
| DATE | Date of<br>Record | MM/DD/YYYY | None | Never | Date of record. |
| DATETIME | Date and time of record | MM/DD/YYYY<br>HH:MM:SS | None | Never | Date and time of record. |
| DAY | Study day<br>number of<br>record | Num | None | Never | Day of study relative to first IP dose. |
| NDAY | Nominal day | Num | day | Never | Schedule visit day of study relative to first IP dose. |
| NOMT | Nominal time<br>since FIRST<br>IP dose | Num | h | Never | Nominal time of study relative to first IP dose. NOMT=0 for first dosing record only. |
| NOMTLD | Nominal time<br>since LAST IP<br>dose prior to<br>sample | Num | h | Never | Nominal time of study relative to last IP dose prior to sample. NOMTLD=0 for dosing records. |
| RTFD | Relative time<br>from FIRST IP<br>dose to<br>current<br>sample time | Num | h | Never | Actual time from FIRST dose of IP. |
| RTLD | Relative time<br>from LAST IP<br>dose prior to<br>sample | Num | h | Never | Actual time from last dose of IP prior to sample. When LABL=DOSE_GSK1325756, RTLD=0. For pre-dose PK sample on Day 7, RTLD is relative to the previous dose. |
| DOSE | Dose amount | Num | mg | Never | DOSE=35. To be entered in all rows for each subject. |

| Variable | Label<br>(Variable<br>description) | Туре | Units | Missing value | Codes/Derivation/Notes |
|---|---|---|---|---|---|
| DRUG | Name of drug | Char | None | Never | DRUG=GSK1325756. To be entered in all rows for each subject. |
| REG | Dosing<br>Regimen | Integer | None | Never | REG=2 for BD. To be entered in all rows for each subject. |
| REGTEXT | Subject dose regimen text | Char | None | Never | REGTXT=BD, text corresponding to code for REG. To be entered in all rows for each subject. |
| ROUT | Route of administration | Integer | None | Never | ROUT=1 for PO. To be entered in all rows for each subject. |
| ROUTTEXT | Subject route of administration text | Char | None | Never | ROUTTEXT=PO, text corresponding to code for ROUT. To be entered in all rows for each subject. |
| CMT | NONMEM<br>Compartment<br>code | Integer | None | Never | CMT=1 for DOSE_GSK1325756 records. CMT=2 for PK_GSK1325756 records. |
| EVID | NONMEM<br>Event ID | Integer | None | Never | EVID=1 for LABL=<br>DOSE_GSK1325756.<br>EVID=0 for LABL=<br>PK_GSK1325756. |
| AMT | NONMEM<br>Amount of<br>drug<br>administered | Num | mg | Never | AMT=0 for LABL= PK_GSK1325756 records. AMT=35 for LABL= DOSE_GSK1325756 records. |
| II | NONMEM<br>Inter-dose<br>interval | Integer | h | Never | II=0 for LABL= PK_GSK1325756. II=12 for LABL= DOSE_GSK1325756, except II=0 for LABL= DOSE_GSK1325756 on Day 1 only. |
| SS | Steady-state data item | Integer | None | Never | SS=0 for LABL= PK_GSK1325756 records. SS=1 for LABL= DOSE_GSK1325756 records, except SS=0 for LABL= DOSE_GSK1325756 records on Day 1 only. |
| RATE | NONMEM<br>Rate of drug<br>infusion | Integer | None | Never | RATE=0 for LABL= PK_GSK1325756 records. RATE=-2 for LABL= DOSE_GSK1325756 records. |

| Variable | Label<br>(Variable<br>description) | Туре | Units | Missing value | Codes/Derivation/Notes |
|---|---|---|---|---|---|
| MDV | NONMEM<br>Missing data<br>value | Integer | None | Never | MDV=1 for LABL= DOSE_GSK1325756 records. MDV=0 for LABL= PK_GSK1325756 records. MDV=1 for LABL= PK_GSK1325756 records < LOQ (NQ). |
| VIS | Visit number | Integer | None | Never | From source data. |
| POP | Population | Integer | None | Never | POP=1, for COPD. To be entered in all rows for each subject. |
| POPTEXT | Subject<br>population<br>text | Char | None | Never | POPTEXT=COPD, text corresponding to code for POP. To be entered in all rows for each subject. |
| СОН | Cohort | Integer | None | Never | COH=1. To be entered in all rows for each subject. |
| AGE | Subject Age | Integer | year | If missing impute with -99 | From source data. To be entered in all rows for each subject. |
| SEX | Subject<br>gender | Integer | None | Never | O=Male, 1=Female To be entered in all rows for each subject. |
| SEXTEXT | Subject<br>gender text | Char | None | Never | Text corresponding to code for SEX, e.g. MALE or FEMALE). To be entered in all rows for each subject. |
| BMI | Baseline Body<br>Mass Index | Num | kg/m² | If missing impute with -99 | Ensure consistent with S&P formula. E.g. Formula: Weight(kg)/(height(m)**2) To be entered in all rows for each subject. |
| BSA | Baseline Body<br>Surface Area | Num | m <sup>2</sup> | If missing impute with -99 | Formula: BSA (m²) = 0.024265 • Height(cm) <sup>0.3964</sup> • Weight(kg) <sup>0.5378</sup> Ensure consistent to with S&P formula. To be entered in all rows for each subject. |
| WT | Baseline<br>Subject<br>weight | Num | kg | If missing impute with -99 | From source data. To be entered in all rows for each subject. |
| HT | Baseline<br>Subject height | Num | m | If missing impute with -99 | From source data. To be entered in all rows for each subject. |
| RACE1 | Subject race code1 | Integer | None | Never | From source data e.g.<br>1=African American / African |

| Variable | Label<br>(Variable<br>description) | Туре | Units | Missing value | Codes/Derivation/Notes |
|---|---|---|---|---|---|
| | | | | | Heritage 2=American Indian or Alaska Native 3=Asian – Central / South Asian Heritage 4=Asian – East Asian Heritage 5=Asian – Japanese Heritage 6=Asian – South East Asian Heritage 7=Asian – Mixed Race 8=Native Hawaiian or other Pacific Islander 9=White – Arabic / North African Heritage 10=White – White / Caucasian / European Heritage 11=White – Mixed Race 12=Mixed Race To be entered in all rows for each subject. |
| RACE1TXT | Subject race text | Char | None | Never | Text corresponding to code for RACE1 To be entered in all rows for each subject. |
| RACE2 | Subject race code2 | Integer | None | Never | 1=East Asian: Asian – East Asian Heritage & Asian – Japanese Heritage 2=White: White – Arabic / North African Heritage White – White / Caucasian / European Heritage 3=African: African American / African Heritage; 4=Other: American Indian or Alaska Native; Asian – Central / South Asian Heritage; Asian – South East Asian Heritage; Asian – Mixed Race; Native Hawaiian or other Pacific Islander; White – Mixed Race & Mixed Race To be entered in all rows for each subject. |
| RACE2TXT | Subject race text | Char | None | Never | Text corresponding to code for RACE2 To be entered in all rows for each subject. |
| ETHN | Subject ethnicity | Num | None | Never | From source data definition. E.g 1=Hispanic or Latino, 2=Non- |

| Variable | Label<br>(Variable<br>description) | Туре | Units | Missing value | Codes/Derivation/Notes |
|---|---|---|---|---|---|
| | | | | | Hispanic To be entered in all rows for each subject. |
| ETHNTEXT | Subject ethnicity text | Char | None | Never | Text corresponding to code for ETHN. To be entered in all rows for each subject. |
| REGN | Region for subject | Num | None | Never | 1 = East Asia (to include Japan,<br>South Korea and Taiwan)<br>2 = Rest of the World (to include<br>all other countries)<br>To be entered in all rows for each<br>subject. |
| SMOK | Subject<br>smoking<br>status | Integer | None | Never | 0=Non-smoker, 1=Smoker,<br>2=Former smoker<br>To be entered in all rows for each<br>subject. Smoking status at<br>baseline. |
| SMOKTEXT | Subject<br>smoking<br>status text | Char | None | Never | Text corresponding to code for SMOK. To be entered in all rows for each subject. |
| CMED1 | Identifier for on-treatment COPD concomitant medication | Num | None | Never | 0 = no concomitant use 1 = intermittent use 2 = continuous use To be entered in all rows for each subject. |
| CMED1TEXT | Subject<br>CMED1 text | Char | None | Never | Text corresponding to code for CMED1. To be entered in all rows for each subject. |
| CRCL | Baseline<br>Creatinine<br>Clearance | Num | mL/min | If missing impute with -99 | From source data. OR Specify appropriate formula e.g. Creatinine Clearance will be calculated based on the Cockcroft-Gault equation. • CrCL (ml/min) = [140 – AGE (in years)]*Weight(kg)*0.85 (for female patients) / [72* Serum Creatinine (micromol/L) * 0.0113 • Delete one as appropriate and ensure consistency with S&P |

| Variable | Label<br>(Variable<br>description) | Туре | Units | Missing value | Codes/Derivation/Notes |
|---|---|---|---|---|---|
| | | | | | formula To be entered in all rows for each subject. |
| CMED2 | Identifier for on-treatment gastric acid reducing concomitant medication | Num | None | Never | 0 = no concomitant use 1 = intermittent use 2 = continuous use To be entered in all rows for each subject. |
| CMED2TEXT | Subject<br>concomitant<br>medication<br>text | Char | None | Never | Text corresponding to code for CMED2. To be entered in all rows for each subject. |
| CMED3 | Identifier for on-treatment gastric acid increasing concomitant medication | Num | None | Never | 0 = no concomitant use 1 = intermittent use 2 = continuous use To be entered in all rows for each subject. |
| CMED3TEXT | Subject<br>concomitant<br>medication<br>text | Char | None | Never | Text corresponding to code for CMED3. To be entered in all rows for each subject. |
| CMED4 | Identifier for on-treatment p-gp inhibitor concomitant medication | Num | None | Never | 0 = no concomitant use 1 = intermittent use 2 = continuous use To be entered in all rows for each subject. |
| CMED4TEXT | Subject<br>CMED4 text | Char | None | Never | Text corresponding to code for CMED4. To be entered in all rows for each subject. |
| CMED5 | Identifier for on-treatment p-gp inducer concomitant medication | Num | None | Never | 0 = no concomitant use 1 = intermittent use 2 = continuous use To be entered in all rows for each subject. |
| CMED5TEXT | Subject<br>concomitant<br>medication<br>text | Char | None | Never | Text corresponding to code for CMED5. To be entered in all rows for each subject. |
| TBIL | Baseline Total bilirubin | Num | Specify | If missing impute with -99 | Baseline defined in the source dataset To be entered in all rows for each subject. |
| TFIB | Baseline<br>Fibrinogen | Num | Specify | If missing impute | Baseline defined in the source dataset |

| Variable | Label<br>(Variable<br>description) | Туре | Units | Missing<br>value | Codes/Derivation/Notes |
|---|---|---|---|---|---|
| | | | | with -99 | To be entered in all rows for each subject. |

**Current Therapies for COPD: CMED1** 

| Long-acting β <sub>2</sub> -agonists (LAE | | |
|---|---|---|
| Formoterol<br>Indacaterol<br>Salmeterol<br>Olodaterol | | |
| Long acting anti-muscarinic a | antagonists (LAMAs) | |
| Tiotropium Aclidinium Bromide Glycopyrronium bromide Umeclidinium | | |
| Long acting combination bro | nchodilators | |
| Albuterol/ipratropium bromide Vilanterol/umeclidinium Olodaterol/tiotropium Indacaterol/glycopyrrolate Formoterol/glycopyrrolate Formoterol/aclidinium | | |
| Methylxanthines | | |
| Theophylline<br>Aminophylline | Bronchodilator effects and claimed anti-inflammatory effects. | Dose-related toxicity including the development of atrial and ventricular arrhythmias and grand mal seizures. |
| Inhaled glucocorticosteroids | | |
| Beclomethasone Budesonide Fluticasone propionate Fluticasone furoate Mometasone | | |

| Inhaled glucocorticosteroids (ICS, in combination with inhaled bronchodilators) | | |
|---|---|---|
| Formoterol/budesonide Salmeterol/Fluticasone propionate Vilanterol/Fluticasone Furoate Formoterol/beclomethasone Formoterol/mometasone | | |
| Inhaled glucocorticosteroids | (ICS, in combination with inh | aled LABA and LAMA) |
| Fluticasone<br>Furoate/Umeclidium/Vilanterol | | |
| Phospodiesterase-4 inhibitors | | |
| Roflumilast | | |
| Antibiotics | | |
| Macrolides (e.g. azithromycin, ervthromycin) | | |

#### CMED2: Gastric acid reducing conmeds

| 0bs | VAR1 | VAR2 |
|---|---|---|
| 1<br>2<br>3<br>4<br>5<br>6<br>7<br>8<br>9<br>10<br>11<br>12<br>13<br>14<br>15<br>16<br>17<br>18<br>19<br>20<br>21<br>22<br>27<br>28<br>29<br>30<br>31<br>32<br>33 | Term Name ESOMEPRAZOLE MAGNESIUM PEPTAZOL (NOS) DOMPERIDONE MALEATE + RABEPRAZOLE SODIUM CLARITHROMYCIN + LANSOPRAZOLE PANTOPRAZOLE ESOMEPRAZOLE DOMPERIDONE + PANTOPRAZOLE ZEGERID (NOS) LANSOPRAZOLE SODIUM ESOMEPRAZOLE STRONTIUM ESOGARD (NOS) OMEPRAZOLE MAGNESIUM ZOLTUM (NOS) TENATOPRAZOLE PRAZOL (NOS) DEXLANSOPRAZOLE DOMPERIDONE + RABEPRAZOLE DOMPERIDONE + RABEPRAZOLE CLARITHROMYCIN + LANSOPRAZOLE + TINIDAZOLE LEVOSULPIRIDE + RABEPRAZOLE SODIUM LEVOSULPIRIDE + RABEPRAZOLE PROTON PUMP INHIBITOR NOS IPP (NOS) OMEPRAZOLE SODIUM PANTOPRAZOLE SODIUM PANTOPRAZOLE SODIUM PANTOPRAZOLE SODIUM POMPERIDONE MAGNESIUM ESOMEPRAZOLE SODIUM POMPERIDONE MALEATE + PANTOPRAZOLE SODIUM PROTONIX (NOS) GASTROZOL (NOS) OMEPRAZOLE + SODIUM BICARBONATE ALIMENTARY TRACT AND METABOLISM; DRUGS FOR LANSOPRAZOLE MOSAPRIDE CITRATE + RABEPRAZOLE SODIUM ESOMEPRAZOLE CITRATE + RABEPRAZOLE SODIUM ESOMEPRAZOLE | 54953101<br>1263201<br>1479301<br>53545101<br>54613401<br>1159002<br>1479304<br>59864501<br>661203<br>59177101<br>1401301<br>53163801<br>53869001<br>53611501<br>53773301<br>53235701<br>54347301<br>54342301<br>54019901<br>661202<br>1263203<br>1479303<br>54543201<br>54724001<br>53827801 |

**NDAY**: For deriving the nominal day which is the planned day, DAY specific information is not available in EXPOSURE dataset. VISIT variable and the time and events table might have to be taken into account to find the exact plan of events.

**NOMT:** It is twice daily dosing with inter-dose interval given to be 12 hours. Therefore, to find the planned time of event since the first dose in hours, again the VISIT variable and time and events will have to be considered.

**NOMTLD**: In case of PK\_GSK1325756 records, the planned time point variable will give the value of this variable for all the post-dose records. For the pre-dose records, this variable will have missing values since there is no fixed time point since the previous dose for pre-dose records.

**RTFD**: The time difference between the first dose of the subject and the current dose (when LABL=DOSE\_GSK1325756) should be calculated in hours. The time difference

between the first dose of the subject and the PK sample collection time (when LABL=PK GSK1325756) should be calculated in hours.

**RTLD**: The latest dose prior to the PK sample collection time will have to be found out and the time difference between that dose and the PK sample collection time will be calculated in hours.

# 12.10. Appendix 10: Abbreviations & Trade Marks

### 12.10.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| AIC | Akaike's Information Criteria |
| A&R | Analysis and Reporting |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| CTR | Clinical Trial Register |
| CV <sub>b</sub> / CV <sub>w</sub> | Coefficient of Variation (Between) / Coefficient of Variation (Within) |
| DBF | Database Freeze |
| DBR | Database Release |
| DOB | Date of Birth |
| DP | Decimal Places |
| eCRF | Electronic Case Record Form |
| EMA | European Medicines Agency |
| FDA | Food and Drug Administration |
| FDAAA | Food and Drug Administration Clinical Results Disclosure Requirements |
| GSK | GlaxoSmithKline |
| IA | Interim Analysis |
| ICH | International Conference on Harmonization |
| IDMC | Independent Data Monitoring Committee |
| IDSL | Integrated Data Standards Library |
| IMMS | International Modules Management System |
| IP | Investigational Product |
| ITT | Intent-To-Treat |
| MMRM | Mixed Model Repeated Measures |
| mITT | Modified Intent to Treat |
| NETs | Neutrophil Extracellular Traps |
| PCI | Potential Clinical Importance |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PK | Pharmacokinetic |
| PP | Per Protocol |
| PopPK | Population PK |
| QĊ | Quality Control |
| QTcF | Frederica's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAP | Reporting & Analysis Plan |
| RAMOS | Randomization & Medication Ordering System |

| Abbreviation | Description |
|--------------|---------------------------------|
| SAC | Statistical Analysis Complete |
| SDSP | Study Data Standardization Plan |
| SDTM | Study Data Tabulation Model |
| SOP | Standard Operation Procedure |
| TA | Therapeutic Area |
| TFL | Tables, Figures & Listings |

### 12.10.2. Trademarks

| Trademarks of the GlaxoSmithKline Group of Companies | |
|------------------------------------------------------|---|
| None | Ī |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| WinNonlin |
| SAS |

### 12.11. Appendix 11: List of Data Displays

### 12.11.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|-------------|-------------|
| Study Population | 1.1 to 1.21 | |
| Efficacy | 2.1 to 2.22 | 2.1 to 2.18 |
| Safety | 3.1 to 3.14 | |
| Pharmacokinetic | 4.1 to 4.2 | 4.1 to 4.6 |
| Section | Listi | ngs |
| ICH Listings | 1 to 30 | |
| Other Listings | 31 to 44 | |

### 12.11.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced by the name of the table or figure and if required example mock-up displays provided in Appendix 12: Example Mock Shells for Data Displays.

#### 12.11.3. Deliverables

| Delivery [Priority] [1] | Description |
|-------------------------|-----------------------------------------|
| SAC [X] | Final Statistical Analysis Complete |
| D | Will be part of the abbreviated dry run |

#### NOTES:

1. Indicates priority (i.e. order) in which displays will be generated for the reporting effort

## 12.11.4. Study Population Tables

| Study | Population Tab | les | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | t Disposition | | | | |
| 1.1. | mITT | ES1 | Summary of Subject Disposition for the Subject Conclusion Record | ICH E3, FDAAA, EudraCT, Use latest screening | SAC [2] |
| 1.2. | mITT | SD1 | Summary of Treatment Status and Reasons for Discontinuation of Study Treatment | ICH E3 | SAC [2] |
| 1.3. | Enrolled | ES6 | Summary of Screening Status and Reasons for Screen Failure | Journal Requirements, Use latest screening. If a subject is rescreened only use final re-screen | SAC [2] |
| 1.4. | Enrolled | NS1 | Summary of Number of Subject by Country and Site ID | EudraCT/Clinical Operations | SAC [2] |
| 1.5. | mITT | NS1 | Summary of Number of Subject by Country and Site ID | EudraCT/Clinical Operations | SAC [2] |
| 1.6. | Primary<br>Completer | NS1 | Summary of Number of Subject by Country and Site ID | EudraCT/Clinical Operations. If the primary completer and mITT population are the same do not recreate | SAC [2] |
| Protoc | ol Deviation | | | | |
| 1.7. | mITT | DV1 | Summary of Important Protocol Deviations | ICH E3 | SAC [2] |
| 1.8. | Enrolled | IE1 | Summary of Inclusion/Exclusion Criteria Deviations for Screen or Run-in failures | | SAC [2] |
| 1.9. | mITT | IE1 | Summary of Inclusion/Exclusion Criteria Deviations for the Modified Intent-to-treat Population | | SAC [2] |

| Study I | Population Tab | les | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Popula | tion Analysed | | | | |
| 1.10. | Enrolled | SP1 | Summary of Study Populations | IDSL Number of participants who were in the Enrolled population, who were randomized, the number in the mITT population. Of those in the mITT, the number and percentage of participants in the primary completer population | SAC [2] |
| Demog | raphic and Bas | seline Characteris | tics | | |
| 1.11. | mITT | DM1 | Summary of Demographic Characteristics | ICH E3, FDAAA, EudraCT | SAC [2] |
| 1.12. | Primary<br>Completer | DM1 | Summary of Demographic Characteristics | ICH E3, FDAAA, EudraCT | SAC [2] |
| 1.13. | Enrolled | DM11 | Summary of Age Ranges | EudraCT | SAC [2] |
| 1.14. | mITT | PD4 | Summary of Screening and Baseline Spirometry Measures | Pre-BD FEV1 (L), Post-BD FEV1 (L), Predicted normal FEV1 (L), Percent predicted normal post-BD FEV1 (%), Percent predicted normal post-BD FEV1: <50%, >=50%, Post-BD FVC (L), Post-BD FEV1/FVC Footnote: Subjects are only supposed to have a Post Sputum Induction FEV1 at baseline if participant was unable to give a sample at Pre-Screening. The pre-screening and screening samples for this measure are combined. | SAC [2] |
| 1.15. | mITT | SU1 | Summary of Smoking History and Smoking Status at Screening | Include smoking status, smoking pack years, cigarettes smoked/day | SAC [2] |
| 1.16. | mITT | DM6 | Summary of Race and Racial Combinations | ICH E3, FDA, FDAAA, EudraCT | SAC [2] |

| Study F | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Prior a | nd Concomitan | t Medications | | | |
| 1.17. | mITT | MH4 | Summary of Current Medical Conditions | ICH E3 | SAC [2] |
| 1.18. | mITT | MH4 | Summary of Past Medical Conditions | ICH E3 | SAC [2] |
| 1.19. | mITT | CM1 | Summary of Concomitant Medications | ICH E3 | SAC [2] |
| 1.20. | mITT | CM1 | Summary of COPD Concomitant Medications Taken Pretreatment | | SAC [2] |
| 1.21. | mITT | CM1 | Summary of COPD Concomitant Medications Taken Post-treatment | | SAC [2] |

# 12.11.5. Efficacy Tables

| Efficacy | r: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| NETs | | | | | |
| 2.1 | Primary<br>Completer | | Summary of Adjusted Mean Change from Baseline of NETs Quantified by Histone-Elastase | | D, SAC [2] |
| 2.2 | Primary<br>Completer | | Summary of Unadjusted Means of NETs | Histone, DNA, and microscopy quantified | D, SAC [1] |
| 2.3 | Modified<br>Primary<br>Completer | | Summary of Unadjusted Means of NETs for the Modified Primary Population | Histone, DNA, and microscopy quantified. This population will only be use if this increases the available sample from the Primary completer population by 20%. | SAC [2] |
| 2.4 | Primary<br>Completer | | Summary Unadjusted Mean Change from Baseline of NETs | Include percent change from baseline | D, SAC [2] |
| 2.5 | Primary<br>Completer | | Summary of the Ratio of Sputum NETs to Sputum Neutrophils | | D, SAC [2] |
| 2.6 | Primary<br>Completer | | Summary of Change from Baseline in the Ratio of Sputum NETs to Sputum Neutrophils | | D, SAC [2] |
| 2.7 | Primary<br>Completer | | Summary of Sputum Neutrophils | | D, SAC [1] |
| 2.8 | Primary<br>Completer | | Summary of Change from Baseline in Sputum Neutrophils | | D, SAC [2] |
| 2.9 | mITT | | Summary of Peripheral Blood Neutrophil NETs Formation | Will be measured by DNA release and microscopy, summarise no PMA and PMA values septately, but include both on the table. Only collected at baseline and day 14 | D, SAC [1] |

| Efficacy | /: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.10 | mITT | | Summary of Change from Baseline in Peripheral Blood<br>Neutrophil NETs Formation | Will be measured by DNA release and Microscopy | D, SAC [2] |
| 2.11 | mITT | | Summary of Sputum Quality | Number of subjects with Insufficient Tissue, Poor Quality, Acceptable, and Good Quality samples see MISPQL variable for quality flag Mean and SD of Squamous epithelial cells. Mean and SD of Viable Leukocytes. | D, SAC [2] |
| 2.12 | Primary<br>Completer | | Summary of Sputum Quality | Number of subjects with Insufficient Tissue, Poor Quality, Acceptable, and Good Quality samples see MISPQL variable for quality flag Mean and SD of Squamous epithelial cells. Mean and SD of Viable Leukocytes. | D, SAC [2] |
| CAT | | | | | |
| 2.13 | mITT | | Summary of Baseline CAT | | SAC [2] |
| Biomar | ker | | | | |
| 2.14 | Primary<br>Completer | | Summary of Change from Baseline Sputum Resistin Levels | | D, SAC [2] |
| 2.15 | Primary<br>Completer | | Summary of Sputum Resistin Levels | | D, SAC [2] |
| 2.16 | Primary<br>Completer | | Summary of Change from Baseline in Sputum Elastase Activity | | D, SAC [2] |
| 2.17 | Primary<br>Completer | | Summary of Sputum Elastase Activity | | D, SAC [2] |

| Efficacy | y: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.18 | mITT | | Summary of Change from Baseline in Ex-Vivo Neutrophil Phagocytosis of Bacteria by Flow Cytometry | | D, SAC [2] |
| 2.19 | mITT | | Summary of Ex-Vivo Neutrophil Phagocytosis of Bacteria by Flow Cytometry | | D, SAC [2] |
| 2.20 | mITT | | Summary of Change from Baseline of Blood Biomarkers | Include plasma fibrinogen and serum C-reactive protein. For values below the LLQ use X/2 | D, SAC [2] |
| 2.21 | mITT | | Summary of Blood Biomarkers | Include plasma fibrinogen and serum C-reactive protein. For values below the LLQ use X/2 | D, SAC [2] |
| Explora | Exploratory | | | | |
| 2.22 | mITT | | Summary of VOCs Variablity | | SAC [2] |

## 12.11.6. Efficacy Figures

| Efficacy | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| NETs | | | | | |
| 2.1 | Primary<br>Completer | | Adjusted Mean (95% CI) Change from Baseline of NETs Quantified by Histone-Elastase | | D, SAC [2] |
| 2.2 | Primary<br>Completer | | Unadjusted Mean and (95% CI) Change from Baseline of NETs Quantified by Histone-Elastase, DNA-Elastase, and Microscopy | Please add text below indicating the number of subjects in each quality category. Percentage change. | D, SAC [2] |

| Efficac | y: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.3 | Modified<br>Primary<br>Completer | | Unadjusted Mean and (95% CI) Change from Baseline of NETs<br>Quantified by Histone-Elastase, DNA-Elastase, and Microscopy<br>for the Modified Primary Population | Please add text below indicating the number of subjects in each quality category. Percentage change. This population will only be use if this increases the available sample from the Primary completer population by 20%. | SAC [2] |
| 2.4 | Primary<br>Completer | | Spaghetti Plot of Change from Baseline of NETs | | D, SAC [2] |
| 2.5 | Primary<br>Completer | | Spaghetti Plot of NETs | | D, SAC [2] |
| 2.6 | Modified<br>Primary<br>Completer | | Spaghetti Plot of NETs for the Modified Primary Population | This population will only be use if this increases the available sample from the Primary completer population by 20%. | SAC [2] |
| 2.7 | Primary<br>Completers | | Spaghetti and Boxplot of Baseline and Day 14 of NETs<br>Quantified by Histone Elastase | | D, SAC [2] |
| 2.8 | Primary<br>Completers | | Spaghetti and Boxplot of Baseline and Day 14 of Neutrophils | | D, SAC [2] |
| 2.9 | mITT | | Spaghetti and Boxplot of Baseline and Day 14 of Peripheral Blood NETs | For no PMA values only. Will be measured by DNA release and microscopy | D, SAC [2] |
| 2.10 | Primary<br>Completer | | Spaghetti Plot of Change from Baseline in the Ratio of Sputum NETs to Sputum Neutrophils | | D, SAC [2] |
| 2.11 | Primary<br>Completer | | Spaghetti Plot of Ratio of Sputum NETs to Sputum Neutrophils | | D, SAC [2] |

| Efficacy: Figures | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.12 | mITT | | Spaghetti Plot of Change from PMA in Peripheral Blood<br>Neutrophil NETs Formation | Facet the plot by the change that occurs on day -1 and on day 14. Will be measure by DNA release and microscopy | D, SAC [2] |
| 2.13 | mITT | | Spaghetti and Boxplot of Peripheral Blood Neutrophil NETs Formation | | D, SAC [2] |
| 2.14 | mITT | | Boxplot of Change from Baseline in Peripheral Blood Neutrophil NETs Formation | For Placebo and treatment | D, SAC [2] |
| 2.15 | Primary<br>Completer | | Spaghetti Plot of Change from Baseline of Sputum Neutrophils | | D, SAC [2] |
| 2.16 | Primary<br>Completer | | Spaghetti Plot of Sputum Neutrophils | | D, SAC [2] |
| Biomar | kers | | | | |
| 2.17 | mITT | | Mean and (95% CI) of Change from Baseline in Ex-Vivo<br>Neutrophil Phagocytosis of Bacteria by Flow Cytometry | | SAC [2] |
| 2.18 | mITT | | Mean and (95% CI) of Change from Baseline of Blood<br>Biomarkers | | SAC [2] |

## 12.11.7. Safety Tables

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events (AEs) | | | | |
| 3.1. | mITT | AE1CP | Summary of All Adverse Events by System Organ Class and Preferred Term | ICH E3 | SAC [2] |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.2. | mITT | AE1 | Summary of Adverse Events of Special Interest | the specific events of interest will be based on the safety review team (SRT) agreements in place at the time of reporting | SAC [2] |
| 3.3. | mITT | AE1CP | Summary All Drug-Related Adverse Events by System Organ Class and Preferred Term | ICH E3 | SAC [2] |
| 3.4. | mITT | AE15 | Summary of Common (>=5%) Non-serious Adverse Events by System Organ Class and Preferred Term (Number of Participant and Occurrences) | FDAAA, EudraCT | SAC [2] |
| Serious | and Other Sig | nificant Adverse l | Events | | |
| 3.5. | mITT | | Summary of Change from Baseline of Spirometry | | SAC [2] |
| 3.6. | mITT | | Summary of Spirometry | | SAC [2] |
| 3.7. | mITT | AE16 | Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Participants and Occurrences) | FDAAA, EudraCT | SAC [2] |
| Labora | tory: Chemistry | / | | | |
| 3.8. | mITT | LB1 | Summary of Chemistry Changes from Baseline | ICH E3 | SAC [2] |
| Labora | tory: Hematolo | gy | | | |
| 3.9. | mITT | LB1 | Summary of Hematology Changes from Baseline | ICH E3 | SAC [2] |
| Labora | tory: Urinalysis | • | | | |
| 3.10. | mITT | LB1 | Summary of Urine Concentration Changes from Baseline | ICH E3 | SAC [2] |
| Labora | tory: Hepatobil | iary (Liver) | | | |
| 3.11. | mITT | LIVER1 | Summary of Liver Monitoring/Stopping Event Reporting | IDSL | SAC [2] |
| ECG | | | | | |
| 3.12. | mITT | EG1 | Summary of ECG Findings | IDSL | SAC [2] |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.13. | mITT | EG2 | Summary of Change from Baseline in ECG Values by Visit | IDSL | SAC [2] |
| Vital Sig | Vital Signs | | | | |
| 3.14. | mITT | VS1 | Summary of Change from Baseline in Vital Signs | ICH E3 | SAC [2] |

### 12.11.8. Pharmacokinetic Tables

| Pharmacokinetic: Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Whole E | Whole Blood Pk | | | | |
| 4.1. | PK | PKCT1 | Summary of Danirixin Whole Blood Pharmacokinetic Concentration-Time Data | | SAC[2] |
| 4.2. | PK | PKPT4 | Summary of Derived Danirixin Whole Blood Pharmacokinetic Parameters | | SAC[2] |

## 12.11.9. Pharmacokinetic Figures

| Pharma | Pharmacokinetic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 4.1. | PK | PKCF1p | Individual Whole Blood Danirixin Concentration-Time Plots by Subject (Linear and Semi-log) | X-axis displays actual relative time Include line for LLQ along with footnote defining LLQ value Include values below LLQ Verlay Day 1 and 14 | SAC [2] |
| 4.2. | PK | PKCF6 | Individual Whole Blood Danirixin Concentration-Time Plots by Day (Linear and Semi-log) | X-axis displays actual relative time Include line for LLQ along with footnote defining LLQ value Include values below LLQ | SAC [2] |
| 4.3. | PK | PKCF4 | Mean (±SD) Whole Blood Danirixin Concentration-Time Plots (Linear and Semi-log) | Include the full SD bars at each time point X-axis displays planned relative time Include line for LLQ along with footnote defining LLQ value | SAC [2] |
| 4.4. | PK | PKCF5 | Median (Range) Whole Blood Danirixin Concentration-Time Plots (Linear and Semi-log) | Include bars for range at each time point X-axis displays planned relative time Include like for LLQ along with footnote defining LLQ value | SAC [2] |

| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| 4.5. | PK | | Scatter plot of Efficacy versus Danirixin Concentration (Trough) | Spumtum Neutrophil Count and<br>Peripheral Blood Neutrophil<br>Count Include Placebo imputed<br>as DNX conc=0ng/mL, include<br>DNX conc=NQ imputed as<br>LLOQ/2, where LLOQ=5ng/mL<br>By Day | SAC [2] |
| 4.6. | PK | | Scatter plot of Safety versus Danirixin Concentration (Trough) | C-reactive Protein (CRP) Include Placebo imputed as DNX conc=0ng/mL, include DNX conc=NQ imputed as LLOQ/2, where LLOQ=5ng/mL By Day | SAC [2] |

## 12.11.10. ICH Listings

| ICH: Lis | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subjec | Disposition | | | , | |
| 1. | Screened | ES7 | Listing of Reasons for Screen Failure | Journal Guidelines | SAC [2] |
| 2. | Enrolled | ES2 | Listing of Reasons for Study Withdrawal | ICH E3 | SAC [2] |
| 3. | mITT | SD2 | Listing of Reasons for Study Treatment Discontinuation | ICH E3 | SAC [2] |
| 4. | mITT | BL1 | Listing of Subjects for Whom the Treatment Blind was Broken | ICH E3 | SAC [2] |
| 5. | mITT | TA1 | Listing of Planned and Actual Treatments | IDSL | SAC [2] |
| Protoco | ol Deviations | | | | |
| 6. | mITT | DV2 | Listing of Important Protocol Deviations | ICH E3 | SAC [2] |
| 7. | mITT | IE3 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | ICH E3, Add a flag if subject got randomized and dosed | SAC [2] |
| Popula | tions Analysed | | | | |
| 8. | Enrolled | SP3 | Listing of Participants Excluded from Any Population | ICH E3 | SAC [2] |
| Demog | raphic and Bas | eline Characteris | tics | | |
| 9. | mITT | DM2 | Listing of Demographic Characteristics | ICH E3 | SAC [2] |
| 10. | mITT | DM9 | Listing of Race | ICH E3 | SAC [2] |
| 11. | mITT | | Listing of Change in Smoking Status from Screening | | SAC [2] |
| Prior a | nd Concomitan | t Medications | | | |
| 12. | mITT | CP_CM3 | Listing of Concomitant Medications | IDSL | SAC [2] |
| Exposu | re and Treatme | ent Compliance | | | |
| 13. | mITT | EX3 | Listing of Exposure Data | ICH E3 | SAC [2] |

| ICH: Lis | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Advers | e Events | | | | |
| 14. | mITT | AE8CP | Listing of All Adverse Events | ICH E3 | SAC [2] |
| 15. | mITT | AE8CP | Listing of Adverse Events of Special Interest | ICH E3 | SAC [2] |
| 16. | Enrolled | AE8CP | Listing of All Adverse Events for Subject not in mITT | ICH E3 | SAC [2] |
| 17. | mITT | AE7 | Listing of Subject Numbers for Individual Adverse Events | ICH E3 | SAC [2] |
| 18. | mITT | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text | IDSL | SAC [2] |
| Serious | and Other Sig | nificant Adverse l | -<br>Events | | |
| 19. | mITT | AE7 | Listing of Adverse Event of Special Interest | the specific events of interest will be based on the safety review team (SRT) agreements in place at the time of reporting | SAC [2] |
| 20. | mITT | AE8CPa | Listing of Fatal Serious Adverse Events | ICH E3 | SAC [2] |
| 21. | mITT | AE8CPa | Listing of Non-Fatal Serious Adverse Events | ICH E3 | SAC [2] |
| 22. | mITT | AE14 | Listing of Reasons for Considering as a Serious Adverse Event | ICH E3 | SAC [2] |
| 23. | mITT | AE8 | Listing of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment | ICH E3 | SAC [2] |
| Hepato | biliary (Liver) | | | | |
| 24. | mITT | MH2 | Listing of Medical Conditions for Subjects with Liver Stopping Events | IDSL | SAC [2] |
| 25. | mITT | SU2 | Listing of Substance Use for Subjects with Liver Stopping Events | IDSL | SAC [2] |

| ICH: Lis | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| All Lab | oratory | | | | • |
| 26. | mITT | LB5 | Listing of All Laboratory Data for Subjects with Any Value of Potential Clinical Importance | ICH E3 | SAC [2] |
| 27. | mITT | LB5 / LB6 | Listing of Laboratory Values | IDSL | SAC [2] |
| 28. | mITT | UR2A | Listing of Urinalysis Data for Subjects with Any Value of Potential Clinical Importance | ICH E3, Use IDSL standard range | SAC [2] |
| ECG | | | | | |
| 29. | mITT | EG3 / EG4 | Listing of ECG Values | IDSL | SAC [2] |
| Vital Si | Vital Signs | | | | |
| 30. | mITT | VS4 / VS5 | Listing of Vital Signs | IDSL | SAC [2] |

# 12.11.11. Non-ICH Listings

| Non-IC | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| NETs | | • | | | |
| 31. | Primary<br>Completer | | Listing of NETs | Include Change from Baseline | SAC [2] |
| 32. | Primary<br>Completer | | Listing of the Ratio of Sputum NETs to Sputum Neutrophils | Include Change from Baseline | SAC [2] |
| 33. | mITT | | Listing of Peripheral Blood Neutrophil NETs Formation | Include Change from Baseline | SAC [2] |
| 34. | Primary<br>Completer | | Listing of Sputum Quality Measures | Quality measure, viability of leukocytes, and Squamous epithelial cells | SAC [2] |
| Spiron | netry | • | | | |
| 35. | mITT | | Listing of Spirometry | Include Change from Baseline | SAC [2] |
| 36. | mITT | | Listing of Baseline CAT | Flag to indicate if they are part of the primary completer population | SAC [2] |
| Explor | atory | | | | |
| 37. | mITT | | Listing of Treatment Adherence | | SAC [2] |
| 38. | mITT | | Listing of VOCs | | SAC [2] |
| Bioma | rker | • | | | |
| 39. | Primary<br>Completer | | Listing of Sputum Resistin | Include Change from Baseline | SAC [2] |
| 40. | Primary<br>Completer | | Listing of Sputum Elastase | Include Change from Baseline | SAC [2] |
| 41. | mITT | | Listing of Ex-Vivo Neutrophil Phagocytosis of Bacteria by Flow Cytometry | Include Change from Baseline | SAC [2] |

| Non-ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 42. | mITT | | Listing of Blood Biomarkers | Include plasma fibrinogen and serum<br>C-reactive protein. Include Change<br>from Baseline | SAC [2] |
| PK | | | | | |
| 43. | PK | PKCL1P | Listing of Danirixin Whole Blood Pharmacokinetic Concentration-Time Data | | SAC [2] |
| 44. | PK | PKPL1P | Listing of Derived Danirixin Whole Blood Pharmacokinetic Parameters | | SAC [2] |

## 12.12. Appendix 12: Example Mock Shells for Data Displays

Available Upon Request